CLINICAL TRIAL: NCT04850001
Title: Investigating the Changes of the Cognition in Asymptomatic Intracranial Stenosis Patients After 1-Year Standard Medical Treatment Without Stenting
Brief Title: Cognitive Decline in Asymptomatic Intracranial Stenosis Patients: A 1-Year Follow-Up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Other Study IDs: AHMU-ICAS-Best
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Magnetic Resonance Imaging; Asymptomatic Intracranial Stenosis; Medical Treatment
Keywords: Magnetic Resonance Imaging; Asymptomatic Intracranial Stenosis patients; Cognitive function; Medical Treatment
MeSH Terms: interventions — Aspirin; Clopidogrel; Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Asymptomatic intracranial stenosis patients who receive standard medical treatment without stenting
  Interventions: Drug: Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin
- Healthy Control: Healthy control are free from intracranial stenosis

INTERVENTIONS:
Drug: Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin — All patients received standard medical management, including dual antiplatelet therapy (aspirin and clopidogrel) for three months with aspirin or clopidogrel monotherapy thereafter and high-dose statin, and treatment of hypertension to guideline targets.
  Groups: Patient Group

SUMMARY:
To investigate the cognitive decline after standard medical treatment without stenting in Asymptomatic Intracranial Stenosis patients and the underlying neural mechanism by fMRI.

DETAILED DESCRIPTION:
All participants underwent a medical evaluation that included routine laboratory studies before and after 1-year standard medical treatment. Upon meeting the inclusion criteria and providing informed consent, each participant will complete a battery measure of neuropsychological tests and Magnetic Resonance imaging scan in multimodalities within 7 days after admission and after 1-year when patients received standard medical treatment at the First Affiliated Hospital of AnHui Medical University. participants were randomly allocated to patient group and the control group.There are about 20 patients and 20 healthy controls in this study.

Firstly, a series of neuropsychological tests were obtained by a trained investigator to assess baseline. Each assessment will involve a set of assessment tools, the memory as the primary outcome measure and various other tasks and questionnaires to measure cognition (including MoCA,MMSE, DS, Stroop test, TMT, VFT), memory (CAVLT), emotion (HAMA-17,HAMD-14), behavioral and psychological symptoms(NPI). All the tests are conducted in two days. The patients had receiving a magnetic resonance imaging scan in multi-modalities.

After 1-year standard medical treatment,the patients participants were interviewed to obtain the same assessment and magnetic resonance imaging scan in multi-modalities as before. Patients are instructed to focus their answers on the past 15 days. The clinical symptom of participants were followed 6 and 12 months after the admission. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intracranial stenosis which was defined as stenosis of 50% or more in Intracranial segment of internal carotid artery and middle cerebral artery (MCA).
* The degree of stenosis was measured by transcranial doppler, computed magnetic resonance angiography (MRA),tomography angiography (CTA) and digital subtraction angiography (DSA).

Exclusion Criteria:

* History of stroke,transient ischemic attack,seizures or unexplained loss of consciousness.
* Organic brain defects on T1 or T2 images.
* Any history or clinical signs of other severe psychiatric illnesses (like major depression,psychosis or obsessive compulsive disorder).
* Implanted pacemaker,medication pump,vagal stimulator,deep brain stimulator. History of substance abuse within the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial stenosis which was defined as stenosis of 50% or more in Intracranial segment of internal carotid artery and middle cerebral artery (MCA) without history of stroke,transient ischemic attack,seizures or unexplained loss of consciousness.The degree of stenosis was measured by transcranial doppler, computed magnetic resonance angiography (MRA),tomography angiography (CTA) and digital subtraction angiography (DSA).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Memory | baseline, 1-year after medical treatment
  The changes in Memory function will constitute the major research outcome measure used to assess response to standard medical treatment.

SECONDARY OUTCOMES:
The changes in MMSE(Mini Mental State Examination) | baseline, 1-year after medical treatment
  The changes in MMSE will constitute the secondary research outcome.The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better. In this study, changes in MMSE scores before and after 1-year medical treatment were used as secondary observations,we suspect that scores would decrease after 1-year medical treatment.
DST (Digital Span Test; Forward and Backward) | baseline, 1-year after medical treatment
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability. There are two types of test: forward(0-14) and backward(0-13).In the forward test, the subjects were asked to retell the the digits immediately after hearing it until they could not be repeated correctly.In backward test, the subjects were asked to repeat a set of numbers in reverse order until they could not be repeated correctly. The length of the last set of Numbers correctly repeated by the subjects was the final score, forward and backward are counted separately. The higher the score, the better. In this study, we suspect that scores would decrease after 1-year medical treatment.
TMT (Trail Making Test) | baseline, 1-year after medical treatment
  The changes in TMT will constitute the secondary research outcome. The Trail Making Test (TMT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.In this study, we suspect that scores would decrease after 1-year medical treatment.
HAMD (Hamilton Depression Scale) | baseline, 1-year after medical treatment
  The changes in HAMD will constitute the secondary research outcome. Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.Higher scores indicate more depressive symptoms. The severity of the disease and the therapeutic effect can be evaluated after treatment. In this study, we suspect that scores would decrease after 1-year medical treatment.
HAMA (Hamilton Anxiety Scale) | baseline, 1-year after medical treatment
  The changes in HAMA will constitute the secondary research outcome. Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959.It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety. The severity of the disease and the therapeutic effect can be evaluated after treatment. In this study, we hoped that scores would decrease after 1-year medical treatment.
MRI measures | baseline, 1-year after medical treatment
  Multimodal magnetic resonance data were acquired, including structural phase magnetic resonance and rest state magnetic resonance, to compare the neuroimaging differences between the patients and healthy control groups before and after 1-year.
changes in Montreal Cognitive Assessment (MoCA) | baseline, 1-year after medical treatment
  MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. We adopted a localized version (Mandarin version，includes 2 alternative versions) in line with the Chinese cultural background.It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score. The final score of the higher the better, and we suspect the subjects' scores will decrease after 1-year medical treatment.
The Stroop color test | baseline, 1-year after medical treatment
  The changes in The Stroop color test will constitute the secondary research outcome measure.The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects. We suspect the participants to spend more time after the medical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No